CLINICAL TRIAL: NCT04055298
Title: Is Self-triage by Patients Using a Symptom-checker Safe?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas Meer (Industry)
Collaborators: Cantonal Hospital of Baden (Unknown)
Responsible Party: Sponsor-Investigator, Andreas Meer, Medical Director, in4medicine AG
Organization: in4medicine AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMASS-Triage_001
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Triage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): The study will be performed at the Walk-in-Clinic (WIC) and Interdisciplinary Emergency Department (ED) of the cantonal hospital of Baden, Switzerland. During their stay at the WIC or ED the patients will be invited to use the triage-symptom-checker SMASS-Triage.
  In this study, the patient's self-triage using a symptom checker will be compared with the urgency assessments conducted by three interdisciplinary panels of physicians (panel A, B and C). In order to appropriately reflect the complex interaction in medical decision-making, which usually leads to a low inter-rater reliability, the cases assessed to be undertriaged by panel A, are subsequently assessed a second time by two panelist of panel B. Cases which are adjudged to be undertriaged by all panelist (panel A and B), are assessed for a risk to health or life by panel C. The risk assessments of panel C will be based on the structured reports generated by the symptom-checker and the discharge summaries of the WIC/ED.
  Interventions: Device: SMASS-Triage

INTERVENTIONS:
Device: SMASS-Triage — SMASS-Triage is a web-based symptom checker developed by In4medicine Ltd. SMASS-Triage is based on a computerized transparent neural network, which was trained with the evidence of more than 1200 studies and the expertise of various panels of specialists in the field of preclinical medical triage. SMASS-Triage provides digitalized questionnaires of 87 frequent reasons of encounters (e.g. fever, cough, abdominal pain) and their associated red flags. The triage-result of SMASS-Triage encompasses the appropriate time-to-treat (T2T) and the adequate point-of-care (PoC).

SUMMARY:
This is a prospective, non-randomized, no placebo-controlled interventional study.

The study aims to assess the safety of the web-based symptom checker SMASS-Triage and its tolerability in terms of incidence of under-triaged self-assessments and the potential risk to be life-threatening or harmful.

The patient's self-triage using a symptom checker will be compared with the urgency assessments conducted sequentially by three interdisciplinary panels of physicians (panel A, B and C). The risk assessments will be based on the structured reports generated by the symptom checker and the discharge summaries of the WIC/ED.

ELIGIBILITY:
Inclusion Criteria:

* All German-, French-, Italian-, English-speaking patients attending the WIC/ED are eligible.
* Informed Consent as documented by signature ( Informed Consent Form)
* Age 18-years and older
* Capable of judgment
* Not under tutelage

Exclusion Criteria:

* Patients with an Emergency Severity Index 1
* Leading complaint of the patient can't be found and assessed with the symptom checker
* Patients not being able to use a tablet-computer
* Patients not speaking German, French, Italian or English
* Minors under the age of 7-years
* Patients incapable of judgment
* Participants under tutelage
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of self-triage assessed to be a hazardous under-triage | Baseline
  The primary endpoint will be the proportion of self-triage and the according confidence interval assessed by the physicians to be a hazardous under-triage.

SECONDARY OUTCOMES:
Proportion of self-triage with an over- or under-triage | Baseline
  Secondary endpoints will be the proportion of self-triage with an over- or under-triaged self-assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meer, MD, MHIM, Principal Investigator — in4medicine Ltd.
Locations (1):
- Cantonal Hospital Baden, Baden, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meer A, Rahm P, Schwendinger M, Vock M, Grunder B, Demurtas J, Rutishauser J. A Symptom-Checker for Adult Patients Visiting an Interdisciplinary Emergency Care Center and the Safety of Patient Self-Triage: Real-Life Prospective Evaluation. J Med Internet Res. 2024 Jun 27;26:e58157. doi: 10.2196/58157. PMID 38809606